CLINICAL TRIAL: NCT06825338
Title: Investigating the Effectiveness of the 'CATCH My Breath' Vaping Prevention Curriculum at Preventing Vaping Initiation Among High School Students in Ontario, Canada
Brief Title: Does the 'CATCH My Breath' Vaping Prevention Program Prevent High School Students in Ontario, Canada From Starting to Vape?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ontario Institute of Technology (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); University of Waterloo (Other); Ontario Agency for Health Protection and Promotion (Other Government); CATCH Global Foundation (Unknown)
Responsible Party: Principal Investigator, Adam Cole, Principal Investigator, University of Ontario Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB-18093; PJT-195799 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: Vaping Behaviors
Keywords: Vaping Prevention; Adolescent; CATCH My Breath; E-cigarette use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: This is a two-arm quasi-experimental study. The study team will recruit schools that will implement the CATCH My Breath vaping prevention curriculum (intervention group). Results will be compared with a separate on-going study of youth health: the COMPASS study (comparison group). Schools recruited into the COMPASS study will not implement the CATCH My Breath vaping prevention curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CATCH My Breath (CMB) (Experimental): CATCH My Breath (CMB) is a school-based vaping prevention curriculum based on best practices from earlier prevention studies that works by fostering social competence and social influence resistance skills. The curriculum design and content targets two key constructs of Social Cognitive Theory: self-efficacy and behavioural capacity (i.e., knowledge and skills). The curriculum provides students with knowledge of why and how to resist vaping. It is delivered through two 60-minute lessons by a trained Public Health Unit presenter. The curriculum lessons provide information about: 1) the physical, mental, and addiction risks associated with vaping, 2) social norms of vaping (e.g., most youth don't vape), 3) media literacy (e.g., how to recognize and decipher marketing of vapes), 4) strategies to resist and avoid vaping, 5)school and provincial policies about vaping. To solidify the content, in-class activities allow students to discuss what they are learning and practice refusal skills.
  Interventions: Other: CATCH My Breath
- Comparison (No Intervention): In Ontario, the current Health and Physical Education curriculum does not include any vaping-specific information, leaving it up to the discretion of educators to decide what to teach and how. The study takes advantage of existing connections to the COMPASS study. The large sample of schools participating in the COMPASS study provides an ideal comparison group, eliminating the need to recruit schools for this condition and reducing costs. The COMPASS study collects information about changes to school programs, policies, and the built environment that may occur over time using the School Policies and Practices survey. This survey is completed annually by a school contact knowledgeable about the school's health-related programs and policies. School contacts are asked whether the school offers any programs that address vaping and tobacco use prevention/cessation. This information will be used to identify schools that have not implemented any vaping/tobacco use programs.

INTERVENTIONS:
Other: CATCH My Breath — CATCH My Breath (CMB) is a school-based vaping prevention curriculum based on best practices from earlier prevention studies that works by fostering social competence and social influence resistance skills. The curriculum design and content targets two key constructs of Social Cognitive Theory: self-efficacy and behavioural capacity (i.e., knowledge and skills). The curriculum provides students with knowledge of why and how to resist vaping. It is delivered through two 60-minute lessons by a trained Public Health Unit presenter. The curriculum lessons provide information about: 1) the physical, mental, and addiction risks associated with vaping, 2) social norms of vaping (e.g., most youth don't vape), 3) media literacy (e.g., how to recognize and decipher marketing of vapes), 4) strategies to resist and avoid vaping, 5)school and provincial policies about vaping. To solidify the content, in-class activities allow students to discuss what they are learning and practice refusal skills.
  Other Names: Vaping prevention program; Vaping prevention curriculum
  Arms: CATCH My Breath (CMB)

SUMMARY:
Vapes (also called e-cigarettes) have increased in popularity among youth in Canada and the United States. Youth who try vaping are at risk of becoming addicted and continuing to vape. To help combat the rise in vaping, there is an urgent need to identify effective ways to prevent youth from experimenting with vaping. Because of the novelty of vapes, there are few school-based programs targeting vaping. This study will investigate whether a vaping prevention curriculum called 'CATCH My Breath' (CMB) prevents high school students from starting to vape.

The investigators will recruit 28 schools in Ontario, Canada into the intervention group, and students at these schools will be presented with the CMB curriculum by Public Health Unit staff. CMB is an evidence-based program that includes two 60-minute lessons that provide students with information about social norms related to vaping, health risks of vaping, media literacy, and in-class activities to practice refusal skills. Students will complete an online survey before being exposed to the curriculum, 3-months later, and 12-months later. The vaping behaviours of these students will be compared to students in a separate study of youth health (i.e., the COMPASS study) who are not given the curriculum.

Evidence from this study will identify whether students exposed to CMB are less likely to start and continue vaping. If effective, CMB can be easily delivered in high schools across Canada in order to reduce the number of students who vape.

DETAILED DESCRIPTION:
Background and Importance: Youth vaping (or e-cigarette use) as increased dramatically among youth populations in Canada and the United States. While the long-term negative effects of vaping are relatively unknown, youth who vape are at risk of becoming addicted to nicotine and continuing to vape. Given the novelty of these devices and their rising popularity among youth, there is an urgent need to identify effective prevention approaches.

Research Aims: The goal of this study is to investigate the effectiveness of the 'CATCH My Breath' (CMB) vaping prevention curriculum at preventing vaping initiation among a cohort of high school students in Ontario, Canada. Specifically, this study will identify whether students exposed to CMB have a lower likelihood of 1) initiating vaping, 2) being susceptible to future vaping, and 3) vaping in the past 30-days at 12-month follow-up, compared to a matched comparison group of students. This study will also investigate whether the effects of the intervention differ according to gender. Methods: Intervention. CMB is a school-based vaping prevention curriculum based on best practices from earlier prevention studies and incorporates theory to foster social competence and social influence resistance skills. It is delivered through two 60-minute lessons delivered by a trained presenter. A pilot study identified components of the program that worked well and what needed to be adapted for a Canadian high school context. Sample. A purposive sample of 28 high schools in Ontario will be recruited and Public Health staff will deliver the curriculum to grade 9 students during Physical Education & Health classes. A matched sample of 28 high schools from a larger pool of schools participating in a separate study of youth health (i.e., the COMPASS study) will be selected as a comparison group. A matched sample of students will be identified from comparison group schools. Data collection & analysis. Students in the intervention group (n=2800) will complete an online survey before exposure to the curriculum and 3-months, and 12-months later to identify changes in vaping knowledge, attitudes, and behaviour. Descriptive analysis of baseline data will produce a profile of demographics and baseline characteristics and identify any imbalances between the intervention and comparison groups that should be accounted for in later analyses. Multilevel regression models will test for intervention effects while controlling for baseline differences through the use of covariates. Expected Outcomes: Evidence from this project will identify whether students exposed to CMB are less likely to start vaping, which will support school-based efforts to prevent vaping initiation and experimentation among youth.

ELIGIBILITY:
School Inclusion Criteria:

* public and private schools in Ontario, English-speaking schools, include students in grades 9 through 12, operate in a standard school/classroom setting (i.e., not a virtual school)

School Exclusion Criteria:

* non-English speaking schools, virtual schools, currently using the CATCH My Breath vaping prevention curriculum

Student Inclusion Criteria:

* enrolled in the class in which the CATCH My Breath curriculum is being delivered

Student Exclusion Criteria:

* not enrolled in the class in which the CATCH My Breath curriculum is being delivered

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5600 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that initiate vaping at 12-month follow-up | baseline and 12-month follow-up
  One validated item will assess ever vaping: "Have you ever tried a vape, also known as an e-cigarette?", with response options 'Yes' and 'No'. This item is consistent with other youth health surveillance studies in Canada and the US and is already present in the COMPASS survey. The question will include a definition of vapes, including examples and images of common brands, to improve the validity of student responses. Students who respond 'No' at baseline will be categorized as 'Never vapers'. Students who never vaped at baseline who respond 'Yes' at follow-up will be categorized as 'Initiated vaping' (outcome of interest), while those who respond 'No' at follow-up will be categorized as 'Did not initiate vaping' (reference group).

SECONDARY OUTCOMES:
Change in susceptibility to future vaping from baseline to 12-month follow-up | baseline and 12-month follow-up
  Three validated items will assess susceptibility to future vaping among students who never vaped: (1) "Have you ever been curious about using a vape?"; (2) "If one of your best friends were to offer you a vape, would you use it?"; and (3) "At any time during the next year do you think you will use a vape?", with response options 'Definitely yes', 'Probably yes', 'Probably not', and 'Definitely not'. Consistent with previous studies, students who never vaped who respond 'definitely not' to all three questions will be considered 'Not susceptible to future vaping', while all others are considered 'Susceptible to future vaping'. The analyses will explore whether intervention group students who are susceptible to future vaping at baseline are more likely to become not susceptible to future vaping at follow-up relative to comparison group students.
Change in number of students reporting past 30-day vaping from baseline to 12-month follow-up | baseline and 12-month follow-up
  One item will assess current (past 30-day) vaping: "On how many of the last 30 days did you use a vape?" (None, 1 day, 2 to 3 days, 4 to 5 days, 6 to 10 days, 11 to 20 days, 21 to 29 days, 30 days [every day]). Students who report vaping at least one day in the last 30 days will be categorized as 'Current vapers', while all others will be categorized as 'Non-current vapers'. The analyses will explore whether intervention group students who currently vape at baseline are more likely to not currently vape at follow-up relative to comparison group students.
Change in knowledge of vaping-related harms from baseline to 3- and 12-month follow-up | baseline, 3-month, and 12-month follow-up
  Students in the intervention group will answer questions assessing knowledge of harms of vaping (9 items related to content delivered in the lessons), perceived positive and negative outcomes of vaping (11 items), subjective norms of vaping (2 items that ask about norms of vaping among their peers), and vaping resistance self-efficacy (4 validated items).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cole, PhD, Principal Investigator — Ontario Tech University

IPD SHARING:
Plan to Share IPD: Yes
Student surveys: Anonymized data for students who have given permission for their data to be used for secondary research purposes and the associated Codebook will be uploaded to Borealis to be stored indefinitely at the end of the project following data analysis and publication. These anonymized data will be available only to specific individuals upon request. The requests will be reviewed and approved by the PI.
  Field Notes Survey: Anonymized data and the associated Codebook will be uploaded to Borealis to be stored indefinitely at the end of the project following data analysis and publication. These anonymized data will be available only to specific individuals upon request. The requests will be reviewed and approved by the PI.
  COMPASS data: Electronic data used for secondary data analysis will not be shared. Those interested in accessing COMPASS data can submit a Data Request Application to the PI of the COMPASS study.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be uploaded to Borealis following data analysis and publication and will be stored indefinitely.
Access Criteria: Anonymized data for students who have given permission for their data to be used for secondary research purposes will be available only to specific individuals upon request. The requests will be reviewed and approved by the PI.